CLINICAL TRIAL: NCT05272813
Title: A Phase I/II Study to Investigate the Efficacy and Safety of MS-553 in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Brief Title: A Study to Investigate the Efficacy and Safety of MS-553 in CLL/SLL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study is terminated due to major protocol revisions.
Sponsor: Shenzhen MingSight Relin Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: MingSight Pharmaceuticals, Inc (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-001-CN
Record Dates: First submitted 2022-02-18; First posted 2022-03-09 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphoid; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: Stage 1 3+3 dose escalation study with expansion to Stage 2
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MS-553 Low Dose (Experimental): MS-553 Low Dose PO BID
  Interventions: Drug: MS-553
- MS-553 Mid Dose-1 (Experimental): MS-553 Mid Dose-1 PO BID
  Interventions: Drug: MS-553
- MS-553 Mid Dose-2 (Experimental): MS-553 Mid Dose-2 PO BID
  Interventions: Drug: MS-553
- MS-553 High Dose (Experimental): MS-553 High Dose PO BID
  Interventions: Drug: MS-553

INTERVENTIONS:
Drug: MS-553 — MS-553

SUMMARY:
This is a Phase I/II, single arm, multi-center, open-label clinical trial of MS-553 in patients with CLL/SLL whose disease relapsed after or was refractory to at lease 1 prior therapy (chemotherapy and/or targeted drug therapy, which must include BTK inhibitor therapy) and who are indicated for treatment per IWCLL2018.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older, male or female.
* Diagnosis of CLL/SLL per IWCLL2018 criteria.
* Patients with relapsed or refractory CLL/SLL who have failed at least 1 prior therapy (chemotherapy and/or targeted drug therapy, which must include BTK inhibitor therapy), are indicated for treatment per IWCLL2018.
* Measurable lesions detected by contrast-enhanced computed tomography (CT): at least one lymph node with a maximum axis of more than 1.5 cm and one measurable vertical dimension.
* WHO/ECOG performance status of 0 to 2.
* Patients with an estimated survival of more than 3 months.

Exclusion Criteria:

* Biopsy-proven and pathologically confirmed current or past transformation to Richter's syndrome.
* Patients with active and uncontrolled autoimmune cytopenia, including autoimmune hemolytic anemia and idiopathic thrombocytopenic purpura.
* Patients who have received any of the following treatments within 14 days prior to the first dose:

  * Major surgery;
  * Glucocorticoids (at a dose equal to or greater than 20 mg/day prednisone or equivalent), unless used by inhalation, topical or intraarticular route, or unless necessary for premedication before and after iodinated contrast dye. After discussion with the Sponsor, steroid therapy at high doses for an extended period may be allowed under the following circumstances:

    1. Treatment of autoimmune hemolysis or autoimmune thrombocytopenia associated with CLL/SLL;
    2. Short-term (within 14 days) use to treat inactive infections of diseases unrelated to CLL/SLL (e.g. arthritis, asthma), which results in acute exacerbation, including steroid dose modifications required for adrenal insufficiency;
  * Cytotoxic chemotherapy or biologic therapy, excepting BCR pathway kinase inhibitors for which a washout of 24 hours prior to the first dose is required.
* Toxicity from prior anti-tumor therapy (chemotherapy, radiotherapy, or biotherapy) did not restore to ≤ Grade 1 (except for alopecia); atrial fibrillation from prior treatment with BTK inhibitors did not restore to ≤ Grade 2.
* Central nervous system (CNS) leukemia or lymphoma, including a history of asymptomatic, previously treated CNS disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities | 28 days

SECONDARY OUTCOMES:
Incidence and severity of adverse events | Assessed throughout the study from the time of first dose of study drug until 30 days after the patient's last dose of study drug or until the event has resolved, stabilized, or an outcome reached, whichever comes first regardless of timing of EoT visit
Overall response rate | up to 24 months
Time to tumor response | During intervention
Disease control rate | During intervention
Progression free survival | During intervention
Overall survival | During intervention
Assessment of minimal residual disease | During intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zhang, MD, Study Director — Shenzhen MingSight Relin Pharmaceuticals Co., Ltd.
Locations (1):
- Peking University People's Hospital, Beijing, Xicheng District, China